CLINICAL TRIAL: NCT00285220
Title: A Prospective, Multi-Center Study to Evaluate the Safety and Effectiveness of Laparoscopic Truncal Vagotomy for the Treatment of Obesity
Brief Title: Safety and Efficacy of Laparoscopic Truncal Vagotomy for the Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: EndoVx, Inc. (Industry); University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00011552
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laparoscopic Truncal Vagotomy

SUMMARY:
This two site study will evaluate the safety and effectiveness of laparoscopic truncal vagotomy for the treatment of obesity with baseline study and 18 month post op follow up.

DETAILED DESCRIPTION:
30 morbidly obese patients evenly enrolled at The University of California San Francisco and at the University of Rochester will be selected for study on a voluntary basis. They will have a BMI of >35 with at least one obesity related comorbidity or a BMI between 40 and 45. Subjects will undergo specific tests of vagal function and baseline metabolic evaluation at baseline.

Thereafter they will undergo a laparoscopic truncal vagotomy. Over 18 months, post operative tests of adequate vagotomy, weight loss, change in body composition and metabolism will be studied.

ELIGIBILITY:
Inclusion Criteria:

* male or female age 25-55
* BMI 35-40 with comorbidity and BMI 40-45 with or without comorbidity
* Stable weight for the last 3 months
* willing to use contraceptives
* motivated to lose weight
* a personal history of at least one professionally supervised 6 month attempt or more than 2 serious attempts to loose weight
* fully ambulatory

Exclusion Criteria:

* sign of prior major abdominal surgery
* history of or signs and /or symptoms of gastro-duodenal ulcer disease
* abnormal vagus nerve testing
* current use of a list of medication

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percent Excess Weight Loss
Absolute Weight Loss
Change in BMI
Change in Percent Body Fat (DEXA)
Change in Percent Body Fat (Impedence)
Change in Lipid Panel (chol, triglycerides, LDL, HDL
Urinary pH
3 day dietary diary
fasting glucose
OGGT with insulin
OGGT with FFA and gut peptides
gastric emptying

SECONDARY OUTCOMES:
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, MD, Principal Investigator — University of California, San Francisco; Marco Pattti, MD, Principal Investigator — University of California, San Francisco; Thad Boss, MD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of California at San Francisco, Dept of Pediatrics, San Francisco, California
  - Strong Health Bariatric Center at Highland Hospital, Rochester, New York